CLINICAL TRIAL: NCT00088946
Title: Parallel, Randomized, Double-Blind, Placebo Controlled Phase II Adjuvant Studies of Erlotinib and Polyphenon E to Prevent the Recurrence and Progression of Tobacco-Related, Superficial Bladder Cancer
Brief Title: Erlotinib and Green Tea Extract (Polyphenon® E) in Preventing Cancer Recurrence in Former Smokers Who Have Undergone Surgery for Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000377681; UCLA-0301091-03
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-08

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage 0 bladder cancer; stage I bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — polyphenon E; Tea; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Polyphenon E plus erlotinib placebo daily for 12 months.
  Interventions: Dietary Supplement: Polyphenon E; Other: Erlotinib placebo
- Arm 2 (Experimental): Erlotinib and Polyphenon E placebo daily for 12 months.
  Interventions: Drug: erlotinib hydrochloride; Other: Polyphenon E
- Arm 3 (Placebo Comparator): Erlotinib placebo and Polyphenon E placebo daily for 12 months.
  Interventions: Other: Erlotinib placebo; Other: Polyphenon E

INTERVENTIONS:
Dietary Supplement: Polyphenon E — 4-200mg capsules PO daily for 12 months
  Other Names: green tea extract
  Arms: Arm 1
Drug: erlotinib hydrochloride — 100 mg PO daily for 12 months
  Other Names: Tarceva
  Arms: Arm 2
Other: Erlotinib placebo — identical to Erlotinib in look and appearance of dosing.
  Arms: Arm 1; Arm 3
Other: Polyphenon E — identical to Polyphenon E in look and appearance of dosing.
  Arms: Arm 2; Arm 3

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Green tea extract (Polyphenon® E) contains certain ingredients that may slow the growth of tumor cells and prevent the recurrence of cancer. Giving erlotinib or green tea extract after surgery may kill any remaining tumor cells and may prevent the recurrence of bladder cancer.

PURPOSE: This randomized phase II trial is studying how well giving erlotinib together with green tea extract works in preventing cancer recurrence in former smokers who have undergone surgery for bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of erlotinib vs green tea extract (Polyphenon® E) vs placebo on the 2-year recurrence rate in former smokers with resected superficial transitional cell carcinoma of the bladder.
* Develop an effective chemopreventative strategy (as an adjunct to standard care) for the medical management of superficial bladder cancer in these patients.

Secondary

* Determine the toxic effects associated with these drugs in these patients.
* Determine a safe and effective chemopreventative dose of erlotinib in these patients.
* Correlate the modulation of 1 or more biomarkers with bladder cancer recurrence and/or progression in patients treated with these drugs.
* Determine the risk of clinical bladder cancer progression in patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (Ta vs T1 vs carcinoma in situ) and participating center. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral erlotinib and oral green tea extract (Polyphenon® E) placebo once daily.
* Arm II: Patients receive oral green tea extract (Polyphenon® E) and oral erlotinib placebo once daily.
* Arm III: Patients receive oral erlotinib placebo and oral green tea extract placebo once daily.

In all arms, treatment continues for 12 months in the absence of disease recurrence or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 330 patients (110 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be former smokers and have ceased smoking at study entry.
* Participants with any previous history of prior cancer diagnosis of Grade 1, 2, or 3, Ta or T1 papillary TCC, or CIS TCC, histologically confirmed, with a newly diagnosed or recurrent tumor within 6 months of accrual who are rendered disease free by standard of care. Patients with Grade 1 papillary tumors must meet at least one of the following additional criteria:

  1. multiple, synchronous tumors (>2)
  2. a single tumor greater than 1 cm in size
* At study entry, patients must have no evidence of disease
* Participants may have been previously treated with intravesical therapy.
* Age>18 years
* Transurethral resection of bladder tumor within 6 months prior to entry on to study
* Participants must have a signed written informed consent
* Agreement with complete abstinence from heterosexual intercourse or with the use of contraception during the treatment phase in women of childbearing potential
* Negative pregnancy test in women of childbearing potential
* Patients must have adequate bone marrow function at study entry (WBC>3000, platelets>100000/mm3, and hemoglobin>10g/dl)
* Patients must have satisfactory renal and hepatic function, defined as plasma creatinine of < 1.5mg/dl, total bilirubin < 1.5, and AST/ALT < 1.5 x the upper limit of normal
* Patients with evidence of obstructive lung disease as the etiology of a low diffusing capacity will still be eligible as long as the chest radiograph does not demonstrate interstitial changes

Exclusion Criteria:

* Prior chemotherapy or radiotherapy
* Prior (within 2 years) or concurrent malignancies, except non-melanomatous skin tumors or carcinoma in situ of the cervix
* Significant medical or psychiatric condition that would make the participant a poor protocol candidate
* TCC greater than or equal to T2 at most recent diagnosis
* Involvement of the upper urinary tract prior to or at the time of initial tumor resection
* Prior treatment with experimental drugs, high dose steroids, or with any other cancer treatment within 4 weeks prior to the first dose of study drug and for the duration of the study
* Positive pregnancy test at any time throughout the course of the study
* Normal consumption of greater than 5 cups of green tea daily
* Participants taking a known CYP 3A4 inducer or food products and medications known to be inhibitors or metabolized by CYP3A4/5 such as erythromycin, ketoconazole, etc. will be excluded since these drugs may be expected to result in altered exposure of Erlotinib
* ECOG performance status > 1
* History of idiopathic pulmonary fibrosis or other interstitial lung disease
* Use of tricyclic antidepressants, including imipramine, dothiepin, and mianserin
* Use within the last 12 months of amiodarone, methotrexate, isoniazid, minocycline, or nitrofurantoin
* History of environmental or occupational metal dust or wood dust exposure
* History of connective tissue disease, including scleroderma, rheumatoid arthritis, Sjogren's Syndrome, or sarcoid
* Significant ophthalmologic abnormalities or patients using contact lenses
* Evidence of interstitial lung disease on chest radiograph
* Patients without obvious interstitial lung disease on chest radiograph will be excluded if they have evidence of parenchymal restrictive lung disease on pulmonary function testing as identified by the following criteria:

  1. Both vital capacity and total lung capacity <80% of predicted value
  2. A diffusing capacity of the lung for carbon monoxide, corrected for hemoglobin, < 75% of predicted value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of a daily oral dose of polyphenon E, erlotinib, or placebo on subjects who are former smokers with a history of superficial bladder cancer on the bladder cancer recurrence rate at two years of any stage or grade of bladder cancer. | 2 years

SECONDARY OUTCOMES:
To address the unmet need in medical management of superficial bladder cancer as an adjunct to standard of care. | 2 years
Assess toxicities associated with daily oral dosing of polyphenon E or erlotinib in subjects at risk for bladder tumor recurrence and to define a safe and effective prevention dose of erlotinib. | 2 years
Correlate the modulation of one or more biomarkers with recurrence of bladder cancer confirming the value as a surrogate endpoint biomarker for bladder cancer recurrence and/or progression. | 2 years
To assess the risk of clinical bladder cancer progression in patients treated with polyphenon E, erlotinib or placebo. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, MD, FACS, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Bladder Cancer Genitourinary Oncology, PC, Phoenix, Arizona
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Santa Monica UCLA Medical Center, Santa Monica, California
  - Mayo Clinic Cancer Center, Rochester, Minnesota